CLINICAL TRIAL: NCT06002152
Title: Superficial Cervical Plexus Block and Quality of Recovery After Thyroidectomy: A Randomized Controlled Trial
Brief Title: Superficial Cervical Plexus Block and Quality of Recovery After Thyroidectomy
Acronym: QoR-SCPB
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2000035991; No NIH funding (Other: 11.09.23)
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Pain
Keywords: Superficial Cervical Plexus Block; Quality of Recovery; Postoperative Pain; Thyroidectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bupivacaine (Experimental): Participants randomized to this arm will receive 10ml of 0.25% bupivacaine on each side of the bilateral block. This will be done after induction of general anesthesia and prior to start of surgery.
  Interventions: Drug: Bupivacaine
- Placebo (Placebo Comparator): Participants randomized to this arm will receive 10ml of saline on each side of the bilateral block. This will be done after induction of general anesthesia and prior to start of surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bupivacaine — After anesthesia induction and prior to the start of surgery, the superficial cervical plexus block will be performed according to standard protocol by an experienced blinded clinician. In this arm, participants will receive 10 milliliters of 0.25% bupivacaine on both sides of their neck for this block. This will be the only intervention administered for purposes of this study.
  Arms: Bupivacaine
Drug: Placebo — After anesthesia induction and prior to the start of surgery, the superficial cervical plexus block will be performed according to standard protocol by an experienced blinded clinician. In this arm, participants will receive 10 milliliters of saline on both sides of their neck for this block. This will be the only intervention administered for purposes of this study.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn whether a superficial cervical plexus block improves quality of recovery after thyroid surgery. Investigators will compare a superficial cervical plexus block with bupivacaine compared to an identical procedure performed saline placebo to see if there is a difference in quality of recovery on the first postoperative day.

The main question to answer is:

• Does a superficial cervical plexus block with bupivacaine compared to placebo improve quality of recovery in patients having thyroid surgery.

Participants will:

* Fill out an initial preoperative survey
* Be randomized to receive a superficial cervical plexus block with bupivacaine or saline placebo while under anesthesia before the surgery starts
* Fill out a survey about recovery on the first day after surgery

DETAILED DESCRIPTION:
Thyroid surgery is associated with mild to moderate post-operative pain, with most patients requiring opioid pain medicine postoperatively. Nerve blocks, such as the superficial cervical plexus block, are an important component of pain control plans. Superficial cervical plexus blocks have been proven to decrease pain and reduce the need for opioid medications in thyroid surgery. However, previous studies were performed before it became common practice to administer a combination of acetaminophen, nonsteroidal anti-inflammatory drugs (NSAIDs), and steroids for thyroid surgery which also help with pain. Whether the superficial cervical plexus block improves pain control and quality of recovery in this context is unknown. This study aims to determine whether the superficial cervical plexus block has an impact on quality of recovery as measured by a survey called the Quality of Recovery-40 (QoR-40).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* American Society of Anesthesiologists Physical Status classification I-III
* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Scheduled for thyroid surgery
* Access to smartphone device or computer with internet connection and has an email address

Exclusion Criteria:

* Non-English speaking
* American Society of Anesthesiologists Physical Status classification > III
* Have an intolerance or contraindication to the medications involved in the study
* Undergoing repeat thyroid surgery
* Undergoing surgery with planned neck dissection
* Plan for admission post-operatively
* Positive pregnancy test on day of surgery (for participants with child-bearing potential)
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery-40 (QoR-40) questionnaire score on postoperative day (POD) 1 | Up to 2 days
  The QoR-40 is a widely used and well validated metric assessing postoperative quality of recovery. It includes 5 subsections investigating the dimensions of 'Emotional State' (9 questions), 'Physical Comfort' (12 questions), 'Psychological Support) (7 questions), 'Physical Independence' (5 questions), and 'Pain' (7 questions) for a total of 40 questions.
  The questions are scored on a 5-point Likert scale. Possible responses range from 1 = 'none of the time' to 5 = 'all of the time'. For negative items, the Likert scale is reversed. The individual scores are summed for the total score which can range from 40 points to 200 points. A higher score indicates better post-operative quality of recovery.
  Participants will be sent an electronic link to the survey via their email. They will complete the surveys privately from their own electronic devices.
  Investigators will then compare the changes in pre-operative vs POD 1 QoR-40 scores between the two groups.

SECONDARY OUTCOMES:
Opioid consumption postoperatively | Up to 2 days
  This outcome will be measured in morphine milligram equivalents. The data will be obtained from electronic medical record (EMR) review. It will be measured from the start of the participant's post-anesthesia care unit (PACU) stay and through POD 1.
Need for rescue analgesia prior to PACU discharge | approximately 4 hours
  This outcome will be measured as "Yes" or "No". The data will be obtained from EMR review from the start of participant's PACU stay to end of participant's PACU stay
Presence of nausea and/or vomiting in the PACU | approximately 4 hours
  This outcome will be measured as "Yes" or "No". The data will be obtained from EMR review. It will be measured from the start of participant's PACU stay to end of participant's PACU stay.
Need for rescue antiemetics in PACU | approximately 4 hours
  This outcome will be measured as "Yes" or "No". The data will be obtained from EMR review. It will be measured from the start of participant's PACU stay to end of participant's PACU stay.
PACU length of stay | approximately 4 hours
  This outcome will be measured in minutes. The data will be obtained from EMR review. It will be measured from the start of participant's PACU stay to end of participant's PACU stay.
Presence of patient reported side effects | up to 2 days
  Participants will self-report any side effects that they experienced post-operatively from the start of their PACU stay and through POD 1.
Patient reported quantity of other modes of analgesia, if any through POD 1 | up to 2 days
  Participants will self-report any other modes of analgesia used post-operatively from the start of PACU stay and through POD 1.

CONTACTS AND LOCATIONS:
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No